CLINICAL TRIAL: NCT00058591
Title: Autologous EBV Specific CTLs for Therapy of Severe Chronic EBV Infection
Brief Title: Treating Severe Chronic Epstein-Barr Virus (EBV) Infection With EBV Specific Cytotoxic T Lymphocytes (CTLs)
Acronym: SCAEBV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Director/Professor, Center for Gene Therapy-Administration, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8216; SCAEBV; NCT00608608 (obsolete NCT alias)
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Epstein-Barr Virus Infections
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Treatment dose levels 1, 2 and 3
  Interventions: Biological: Intravenous injection of EBV specific CTLS

INTERVENTIONS:
Biological: Intravenous injection of EBV specific CTLS — The dose levels for this study are as follows:
  Level Dose
  1. 2 x 107 CTLs/m2
  2. 5 x 107 CTLs/m2
  3. 1 x 108 CTLs/m2
  If patients have a clinical response to the first infusion defined by an improvement in the fatigue score or resolution of clinical abnormalities such as lymphadenopathy or an improvement in laboratory parameters such as a decrease in VCA titer or reduction in free EBV DNA they will be eligible to receive up to 3 additional injections of CTLs at the original dose at 3 monthly intervals.

SUMMARY:
Severe chronic active Epstein-Barr virus (SCAEBV) is a rare Epstein-Barr virus (EBV or commonly known as mono or the kissing disease) associated disorder. This disorder may cause chronic tiredness and fevers and sometimes be complicated by life threatening problems such as multi-organ failure, chronic (ongoing) pneumonia, and lymphoproliferative diseases (diseases involving the lymph nodes which could eventually show up as leukemia or a tumor). The reasons for the body's inability to control the EBV infection are still unknown and no effective treatment is currently available.

This research study uses Epstein-Barr virus (EBV) specific cytotoxic T lymphocytes (CTLs). We want to see if we can grow special white blood cells, called T cells, that have been trained to kill EBV infected cells in the laboratory and see if these cells may help control the EBV infection when given back to the patient.

The purpose of this study is to find the largest safe dose of EBV specific CTLs, to learn what the side effects are, and to see whether this therapy might help the body fight off the SCAEBV infection.

DETAILED DESCRIPTION:
Ten to sixty ml (2-12 teaspoons) of blood will be collected from the patient which we use to grow the T cells. These T cells are then stimulated with EBV infected cells (which have been treated with radiation so that they cannot grow). This stimulation trains the T cells to kill EBV infected cells. We then test the T cells to make sure that they kill the EBV infected cells.

Therapy can take place in one of the specifically designated outpatient clinics so hospital admission is not required. First, patients will be given doses of Tylenol (for any aches/pains) and Benadryl (for any minor allergic reactions such as itching/rash). Next, the T cells will be injected into a vein over a 10 minute period. Patients will be closely watched for any side effects.

If a patient shows some response to the treatment they may receive up to three additional T cell injections at three month intervals. Patients will need to be seen every other week in the clinic for six weeks after the injection. Following that, patients will either be seen in the clinic or contacted by one of the research staff working on this study, once a month for one year.

To learn more about the way the T cells are working and how long they last in the body, an extra 40 mls(8 teaspoonfuls) of blood will be taken at these visits. Additionally, 3 mls (1/2 teaspoonful) of blood will be taken prior to the infusion and monthly thereafter to conduct a CBC (a test to look at the components of the blood).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have severe chronic EBV infection as manifested by 6 months of symptoms Either elevated peripheral blood EBV DNA (>4000 genomes per ug PBMC DNA) or free EBV DNA in serum or CSF or VCA antibody titer > 1/640
* Seronegative for HIV
* Not on investigational agents in the last 4 weeks
* Signed informed consent obtained from patient/guardian
* CTLs available
* Performance status; Karnofsky >60
* Creatinine < 3X normal
* Bilirubin < 5X normal
* Normal electrolytes, calcium, phosphorus, nutritional status
* Females with child-bearing potential must utilize effective birth control.

Exclusion Criteria:

* Patients with a severe intercurrent infection
* Patients that recently received high dose steroids within the last week or other immunosuppressive drugs within a week (or longer as indicated by the half life of the agent)
* Patients with life expectancy of less than 6 weeks
* Pregnant or lactating females

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2000-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to determine the safety of intravenous injections of autologous EBV specific cytotoxic T cell lines in individuals with severe chronic EBV infection | 1 yr

SECONDARY OUTCOMES:
determine antiviral and immunological efficacy of intravenous injections of CTLs in these patients | 1 yr
assess the clinical effects of these injections | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Center for Cell and Gene Therapy, Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas